CLINICAL TRIAL: NCT02305914
Title: A Large Sample Follow-up Study of Long-term Complications of Acute Pancreatitis
Brief Title: Follow-up Study of Complications of Acute Pancreatitis
Acronym: FSCAP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Lingyu Luo, Physician-in-charge, The First Affiliated Hospital of Nanchang University
Other Study IDs: FirstNanchangU
Record Dates: First submitted 2014-11-14; First posted 2014-12-03 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2014-11

CONDITIONS: Pancreatitis; Pancreatic Neoplasms; Metabolic Diseases; Hypertension, Portal; Respiratory Failure; Quality of Life
Keywords: acute pancreatitis; chronic pancreatitis; pancreatic cancer; pancreatic disease-associated portal hypertension; autoimmune pancreatitis; PaO2/FiO2<200; diabetes mellitus; blood lipid; local complications; quality of life
MeSH Terms: conditions — Pancreatitis; Pancreatic Neoplasms; Metabolic Diseases; Hypertension, Portal; Respiratory Insufficiency; Pancreatitis, Chronic; Autoimmune Pancreatitis; Diabetes Mellitus

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — Blood sample faeces sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- follow-up visit: Patients who come for follow-up visit will fill in the questionnaire and undergo regular laboratory examination such as liver function test and CRP,faecal elastase-1 as well as CT scanning.Additionally,blood sample of every patient will be collected and sent to the Lab for storage and further experimented.

SUMMARY:
This is a follow-up study focusing on long-term complications of acute pancreatitis. The primary purposes include: 1. To assess the incidence of type 2 diabetes mellitus（2-DM）,impaired glucose tolerance, metabolic abnormalities of blood lipids after acute pancreatitis. 2. To observe the possible long-term clinical outcomes after acute pancreatitis attack, which may include: chronic pancreatitis, pancreatic cancer, pancreatogenic portal hypertension, autoimmune pancreatitis et al. 3. To evaluate the long-term influence of acute lung injury(PaO2/FiO2<200,FiO2 means fraction of inspiration O2) in AP patients during ICU stay on life qualities of the patients; 4. To observe the prognosis of the local complications of acute pancreatitis(AP) patients; it might be helpful to find the most effective and targeted interventions aiming at different phases after AP attack.

DETAILED DESCRIPTION:
Currently，follow-up study is limited on glucose intolerance and life quality assessment. However, it has been shown that AP is associated to some extent with other diseases such as chronic pancreatitis, pancreatic cancer, pancreatogenic portal hypertension and autoimmune pancreatitis; In addition, for patients who have severe lung injury following AP, especially with PaO2/FiO2<200 during ICU stay, the long term prognosis remains unclear. Thus, a large sample follow-up study is essential for elucidating the possible long-term complications.

Prior to follow up study, the investigators performed baseline analysis of AP patient data from the database of the First Affiliated Hospital of Nanchang University. It is estimated that 1300 patients will be interviewed over telephone and 600 patients in the outpatient department. The content of the follow-up includes: questionnaire (the MOS[medical outcome study] item short from health survey, SF[short form]-36) ; lab testing(complete blood count, blood chemistry such as liver and kidney function, C-reaction protein(CRP), AMY, fasting blood-glucose，1 and 2 hour postprandial blood glucose,C-peptide, blood lipids, FE-1) and CT scan. For patients who have severe lung injuries during ICU stay, pulmonary function test, Blood gas analysis and chest CT will be performed. After screening, the patients with chronic pancreatitis(CP), pancreatic cancer(PC), post Pancreatogenic portal hypertension（PPH） or autoimmune pancreatitis(AIP）will be hospitalized for further therapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute pancreatitis from our hospital
* Must be signed the informed consent

Exclusion Criteria:

* Failed to complete the questionnaire survey and the follow-up examination

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinical diagnosis of acute pancreatitis from the First Affiliated Hospital of Nanchang University from 2005 and 2014,with a follow-up interval of at least 1 year.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-01 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
change in glucose | An expected duration which estimated to be average of 4.2 years
  Fasting blood-glucose，1 and 2 hour postprandial blood glucose will be performed in order to diagnose patients with impaired fasting glucose, impaired glucose tolerance and diabetes according to 2006 World Health organization diagnostic criteria.
Change in C-Peptide | An expected duration which estimated to be average of 4.2 years
  Fasting C-Peptide，1 and 2 hour postprandial C-Peptide will be performed in order to test pancreatic β-cell function.
Change in blood liquid | An expected duration which estimated to be average of 4.2 years
  Blood liquid(triglyceride, cholesterol, low density lipoprotein and high-density lipoprotein) will be tested aiming at evaluating blood liquid metabolism.
Change in the Levels of fecal elastase-1 | An expected duration which estimated to be average of 4.2 years
  Fecal elastase-1(FE-1) were used to evaluate exocrine function. Exocrine insufficiency is defines as FE-1 level less than 200 Kg/g

SECONDARY OUTCOMES:
Abdomen CT | An expected duration which estimated to be average of 4.2 years
  Abdomen CT(preferably enhancing) will be performed for each patient. If CT provides images of pancreatic calcification, pseudocyst, and irregular dilations of the pancreatic ducts, irregular borderline or shape of pancreas and so on, then chronic pancreatitis is suspected; If CT provides images of mass, then further examination should be performed to exclude pancreatic cancer. If CT shows diffuse enlargement with delayed enhancement(sometimes associated with rim-like enhancement) and segmental/focal enlargement with delayed enhancement, then autoimmune pancreatitis should be suspected. Pancreatic disease-associated portal hypertension is suspected if CT indicates splenomegaly and/or portal vein becomes broader.Furthermore, local complications of acute pancreatitis(pancreatic pseudocyst, and walled-off necrosis )according to 2012 revision of the Atlanta classification and definition by international consensus are also observed.
the MOS item short from health survey, SF-36 | An expected duration which estimated to be average of 4.2 years
  To make health study of acute pancreatitis patients through SF-36 for patients fpr patients with PaO2/FiO2<200.
outpatient clinic and phone questionnaire | An expected duration which estimated to be average of 4.2 years

CONTACTS AND LOCATIONS:
Overall Officials: Nonghua Lv, MD, Study Chair — The First Affiliated Hospital of Nanchang University
Locations (1):
- the First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

REFERENCES:
- [Background] McNabb-Baltar J, Ravi P, Isabwe GA, Suleiman SL, Yaghoobi M, Trinh QD, Banks PA. A population-based assessment of the burden of acute pancreatitis in the United States. Pancreas. 2014 Jul;43(5):687-91. doi: 10.1097/MPA.0000000000000123. PMID 24694835
- [Background] Peery AF, Dellon ES, Lund J, Crockett SD, McGowan CE, Bulsiewicz WJ, Gangarosa LM, Thiny MT, Stizenberg K, Morgan DR, Ringel Y, Kim HP, DiBonaventura MD, Carroll CF, Allen JK, Cook SF, Sandler RS, Kappelman MD, Shaheen NJ. Burden of gastrointestinal disease in the United States: 2012 update. Gastroenterology. 2012 Nov;143(5):1179-1187.e3. doi: 10.1053/j.gastro.2012.08.002. Epub 2012 Aug 8. PMID 22885331
- [Background] Papachristou GI, Clermont G, Sharma A, Yadav D, Whitcomb DC. Risk and markers of severe acute pancreatitis. Gastroenterol Clin North Am. 2007 Jun;36(2):277-96, viii. doi: 10.1016/j.gtc.2007.03.003. PMID 17533079
- [Background] Urushihara H, Taketsuna M, Liu Y, Oda E, Nakamura M, Nishiuma S, Maeda R. Increased risk of acute pancreatitis in patients with type 2 diabetes: an observational study using a Japanese hospital database. PLoS One. 2012;7(12):e53224. doi: 10.1371/journal.pone.0053224. Epub 2012 Dec 27. PMID 23300896
- [Background] Xue Y, Sheng Y, Dai H, Cao H, Liu Z, Li Z. Risk of development of acute pancreatitis with pre-existing diabetes: a meta-analysis. Eur J Gastroenterol Hepatol. 2012 Sep;24(9):1092-8. doi: 10.1097/MEG.0b013e328355a487. PMID 22668873
- [Background] Wu D, Xu Y, Zeng Y, Wang X. Endocrine pancreatic function changes after acute pancreatitis. Pancreas. 2011 Oct;40(7):1006-11. doi: 10.1097/MPA.0b013e31821fde3f. PMID 21705952
- [Background] Boreham B, Ammori BJ. A prospective evaluation of pancreatic exocrine function in patients with acute pancreatitis: correlation with extent of necrosis and pancreatic endocrine insufficiency. Pancreatology. 2003;3(4):303-8. doi: 10.1159/000071768. PMID 12890992
- [Background] Das SL, Singh PP, Phillips AR, Murphy R, Windsor JA, Petrov MS. Newly diagnosed diabetes mellitus after acute pancreatitis: a systematic review and meta-analysis. Gut. 2014 May;63(5):818-31. doi: 10.1136/gutjnl-2013-305062. Epub 2013 Aug 8. PMID 23929695
- [Background] Khan AS, Latif SU, Eloubeidi MA. Controversies in the etiologies of acute pancreatitis. JOP. 2010 Nov 9;11(6):545-52. No abstract available. PMID 21068485
- [Background] Anderson F, Thomson SR, Clarke DL, Buccimazza I. Dyslipidaemic pancreatitis clinical assessment and analysis of disease severity and outcomes. Pancreatology. 2009;9(3):252-7. doi: 10.1159/000212091. Epub 2009 Apr 29. PMID 19407479
- [Background] Deng LH, Xue P, Xia Q, Yang XN, Wan MH. Effect of admission hypertriglyceridemia on the episodes of severe acute pancreatitis. World J Gastroenterol. 2008 Jul 28;14(28):4558-61. doi: 10.3748/wjg.14.4558. PMID 18680239
- [Background] Garg PK, Tandon RK. Survey on chronic pancreatitis in the Asia-Pacific region. J Gastroenterol Hepatol. 2004 Sep;19(9):998-1004. doi: 10.1111/j.1440-1746.2004.03426.x. PMID 15304116
- [Background] Levy P, Barthet M, Mollard BR, Amouretti M, Marion-Audibert AM, Dyard F. Estimation of the prevalence and incidence of chronic pancreatitis and its complications. Gastroenterol Clin Biol. 2006 Jun-Jul;30(6-7):838-44. doi: 10.1016/s0399-8320(06)73330-9. PMID 16885867
- [Background] Tandon RK, Sato N, Garg PK; Consensus Study Group. Chronic pancreatitis: Asia-Pacific consensus report. J Gastroenterol Hepatol. 2002 Apr;17(4):508-18. doi: 10.1046/j.1440-1746.2002.02762.x. PMID 11982735
- [Background] Wang LW, Li ZS, Li SD, Jin ZD, Zou DW, Chen F. Prevalence and clinical features of chronic pancreatitis in China: a retrospective multicenter analysis over 10 years. Pancreas. 2009 Apr;38(3):248-54. doi: 10.1097/MPA.0b013e31818f6ac1. PMID 19034057
- [Background] Rickels MR, Bellin M, Toledo FG, Robertson RP, Andersen DK, Chari ST, Brand R, Frulloni L, Anderson MA, Whitcomb DC; PancreasFest Recommendation Conference Participants. Detection, evaluation and treatment of diabetes mellitus in chronic pancreatitis: recommendations from PancreasFest 2012. Pancreatology. 2013 Jul-Aug;13(4):336-42. doi: 10.1016/j.pan.2013.05.002. Epub 2013 May 17. PMID 23890130
- [Background] Bang UC, Benfield T, Hyldstrup L, Bendtsen F, Beck Jensen JE. Mortality, cancer, and comorbidities associated with chronic pancreatitis: a Danish nationwide matched-cohort study. Gastroenterology. 2014 Apr;146(4):989-94. doi: 10.1053/j.gastro.2013.12.033. Epub 2013 Dec 31. PMID 24389306
- [Background] Shimosegawa T, Chari ST, Frulloni L, Kamisawa T, Kawa S, Mino-Kenudson M, Kim MH, Kloppel G, Lerch MM, Lohr M, Notohara K, Okazaki K, Schneider A, Zhang L; International Association of Pancreatology. International consensus diagnostic criteria for autoimmune pancreatitis: guidelines of the International Association of Pancreatology. Pancreas. 2011 Apr;40(3):352-8. doi: 10.1097/MPA.0b013e3182142fd2. PMID 21412117
- [Background] Ikeura T, Miyoshi H, Uchida K, Fukui T, Shimatani M, Fukui Y, Sumimoto K, Matsushita M, Takaoka M, Okazaki K. Relationship between autoimmune pancreatitis and pancreatic cancer: a single-center experience. Pancreatology. 2014 Sep-Oct;14(5):373-9. doi: 10.1016/j.pan.2014.04.029. Epub 2014 Apr 21. PMID 25278307
- [Background] Duell EJ, Lucenteforte E, Olson SH, Bracci PM, Li D, Risch HA, Silverman DT, Ji BT, Gallinger S, Holly EA, Fontham EH, Maisonneuve P, Bueno-de-Mesquita HB, Ghadirian P, Kurtz RC, Ludwig E, Yu H, Lowenfels AB, Seminara D, Petersen GM, La Vecchia C, Boffetta P. Pancreatitis and pancreatic cancer risk: a pooled analysis in the International Pancreatic Cancer Case-Control Consortium (PanC4). Ann Oncol. 2012 Nov;23(11):2964-2970. doi: 10.1093/annonc/mds140. Epub 2012 Jul 5. PMID 22767586
- [Background] Tong GX, Geng QQ, Chai J, Cheng J, Chen PL, Liang H, Shen XR, Wang DB. Association between pancreatitis and subsequent risk of pancreatic cancer: a systematic review of epidemiological studies. Asian Pac J Cancer Prev. 2014;15(12):5029-34. doi: 10.7314/apjcp.2014.15.12.5029. PMID 24998582
- [Background] Koklu S, Yuksel O, Arhan M, Coban S, Basar O, Yolcu OF, Ucar E, Ibis M, Ertugrul I, Sahin B. Report of 24 left-sided portal hypertension cases: a single-center prospective cohort study. Dig Dis Sci. 2005 May;50(5):976-82. doi: 10.1007/s10620-005-2674-x. PMID 15906778
- [Background] Xu LS, Liu JH, Lin P, Huang KH, Chen QK, Chen YT, Zhu ZH. [Clinical features of panereatic disease-associated portal hypertension]. Nan Fang Yi Ke Da Xue Xue Bao. 2010 Jun;30(6):1234-6. Chinese. PMID 20584644
- [Background] Herridge MS, Tansey CM, Matte A, Tomlinson G, Diaz-Granados N, Cooper A, Guest CB, Mazer CD, Mehta S, Stewart TE, Kudlow P, Cook D, Slutsky AS, Cheung AM; Canadian Critical Care Trials Group. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med. 2011 Apr 7;364(14):1293-304. doi: 10.1056/NEJMoa1011802. PMID 21470008
- See also: the First Affiliated Hospital of Nanchang University — http://www.cdyfy.com/